CLINICAL TRIAL: NCT01467206
Title: Life After STroke - the LAST Study. A Norwegian Multi Centre Randomized Controlled Trial
Brief Title: Life After STroke - the LAST Study
Acronym: LAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Asker & Baerum Hospital (Other); The Research Council of Norway (Other); Helse Midt-Norge (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 205309/H10
Record Dates: First submitted 2011-10-31; First posted 2011-11-08 (Estimated); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Cerebral Infarction; Cerebral Hemorrhage
Keywords: Stroke; Physiotherapy; Motor training; Rehabilitation
MeSH Terms: conditions — Cerebral Infarction; Cerebral Hemorrhage; Stroke | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Long term follow up program (Experimental)
  Interventions: Behavioral: Long term follow up by a coordinating physiotherapist
- Standard care (Active Comparator)
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Behavioral: Long term follow up by a coordinating physiotherapist — Monthly meetings with an coordinating physiotherapist who motivate and encourage the patient to do 60 minutes of weekly exercise and 30 minutes of daily physical activity
  Arms: Long term follow up program
Behavioral: Standard care — Standard care as it is given to all stoke patients after stroke
  Arms: Standard care

SUMMARY:
The LAST study is a Norwegian multi site randomised controlled trial that intends to assess the effect of a long term follow up program after stroke. The program consists of a coordinating physiotherapist who will encourage and motivate included patients to perform at least 60 minutes of intensive motor training every week and 30 minutes of physical activity every day for 18 months after inclusion. The primary hypothesis is that patients receiving a long term follow up program after stroke will have better motor function at end of follow up than patients receiving standard care. A total of 390 home dwelling stroke patients living in the municipality of Trondheim, Asker and Bærum will be included at the out-patient clinic at St. Olavs Hospital or Bærum Hospital three months after their stroke. Included patients will be randomised to an intervention group receiving the long term follow up program or to a control group receiving standard care. Motor function, mental health and physical functioning in daily life will be assessed at inclusion and 18 months later. The LAST study is funded by the Norwegian Research Council, the Norwegian University of Science and Technology and the Central Norway Regional Health Authority and will conclude at the end of 2015.

DETAILED DESCRIPTION:
Supplement to the Life After Stroke - the LAST study ClinicalTrials.gov ID: NCT01467206

Changes in the planned statistical analysis, November 9, 2015 The original plan for statistical analysis was published in; Askim T, Langhammer B, Ihle-Hansen H, Magnussen J, Engstad T, Indredavik B. A Long-Term Follow-Up Programme for Maintenance of Motor Function after Stroke: Protocol of the life after Stroke-The LAST Study. Stroke Res Treat. 2012;2012:392101. doi: 10.1155/2012/392101. Epub 2012 Nov 22.

Original plan for statistical analysis Reporting will follow the CONSORT statement for parallel group randomized trials [40]. Descriptive statistics will be performed in order to present the population and the characteristic of the two groups. All analyses will be analysed as intention-to-treat analysis according to the CONSORT instructions. Analysis of covariance (ANCOVA) will be used to study differences between groups according to the primary endpoint, motor assessment scale at 18 months after inclusion. The ANCOVA model will include stroke severity, age, pre stroke disability, treatment group, and motor function at baseline as covariates. Mann-Whitney U test will be used for secondary data not being normal distributed. In all analyses we will control for potential confounding factors, investigate effect modifications, and present both unadjusted and adjusted effects with 95% confidence intervals.

Subanalysis will be performed according to the stratification variables (stroke severity, age above 80 and recruitment site) to explore trends within subgroups of patients.

Revised plan for statistical analysis Reporting will follow the CONSORT statement for parallel group randomized trials [40]. Descriptive statistics will be performed in order to present the population and the characteristic of the two groups. All analyses will be analysed as intention-to-treat analysis according to the CONSORT instructions. Analysis of covariance (ANCOVA) will be used to study differences between groups according to the primary endpoint, motor assessment scale at 18 months after inclusion. The ANCOVA model will include stroke severity, age, pre stroke disability, treatment group, and motor function at baseline as covariates. Similar ANCOVA analyses will be used for the relevant secondary endpoints. Mann-Whitney U test will be used for secondary data not being normal distributed.

Subanalysis will be performed according to the stratification variables (stroke severity, age above 80 and recruitment site), gender, and cognitive status (Mini Mental State below 25), to explore trends within subgroups of patients.

Missing values will be handled using single imputation (typically for items on instrument scales), or by multiple imputation, as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stroke according to WHO's definition of stroke
* Living in the city of Trondheim or the municipalities of Asker or Bærum
* Included 2.5 - 4 months after stroke
* Modified Rankin Scale 0 - 4
* Living at home
* Mini Mental State Examination > 20 or > 16 if aphasia
* Provide informed consent

Exclusion Criteria:

* Are already included in the study
* Are included in other experimental studies
* Unstable coronary function
* Uncompensated heartfailure
* Other diseases that make it difficult to complete the intervention

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Motor Assessment Scale | 18 months after inclusion
  A measure of over all motor function

SECONDARY OUTCOMES:
Barthel Index | 18 months follow up
  A measure of activities of daily living
Modified Rankin Scale | 18 months follow up
  A measure of dependency/independency
Berg Balance Scale | 18 months follow up
  A measure of balance related to basic movement tasks
Timed Up and Go | 18 months follow up
  A measure of balance related to transfer and walking
Sit to stand test | 18 months follow up
  A measure of dynamic muscle strength according to a sit to stand task
Six minute walk test | 18 months follow up
  A measure of endurance
Stroke Impact Scale | 18 months follow up
  A measure of health related quality of life after stroke
EuroQol 5D | 18 months follow up
  A simple measure of health related quality of life for the general population
Fatigue Severity Scale | 18 months follow up
  A measure of the presence of fatigue
One simple question on fatigue from the HUNT3 questionnaire | 18 months follow up
  A simple question used to assess tiredness in teh general Norwegian population
Hospital Anxiety and Depression Scale | 18 months follow up
  A measure of anxiety and depression
Mini Mental State Examination | 18 months follow up
  A measure of cognitive function
Montreal Cognitive Assessment | 18 months follow up
  A measure of cognitive function related to vascular dementia
falls | 6, 12 and 18 months
  Serious falls will be recorded from the patients hospital records
Readmission to hospital | 6, 12 and 18 months
  Number of readmissions to hospital will be recorded from the patients medical records
Death | 6, 12 and 18 months
  Information about death will be collected from the Norwegain Death Registry
Fractures | 6, 12 and 18 months
  Information about fractures during follow up will be collected from the patients medical records
Cardiovascular events | 6, 12 and 18 months
  Information about any cardiovascular events will be collected from the patients medical record
Cerebrovascular events | 6, 12 and 18 months
  Information about any cerebrovascular events during follow up will be collected from teh patient's medical records
International Physical Activity Questionnaire | 6, 12 and 18 months
  A measure of physical activity over the last week
Physical activity assessed by ActivPAL sensor system | 6, 12 and 18 months
  A sensor system to assess the amount of physical activity during a 4-7 day period
Three simple questions on physical activity from the HUNT questionnaire | 18 months
  A simple measure of physical activity
Health costs | 6, 12 and 18 months
  Information about the use of health services will be collected by reviewing the patients' hospital records and records in primary health care system.
National Institutes of Health Stroke Scale | 18 months follow up
  A measure of stroke severity
Modified Ashworth Scale | 18 months follow up
  A measure to rate the degree of spasticity after stroke
Gait speed | 18 months follow up
  A simple measure of maximum gait speed across a 10 metres distance
Trailmaking test A and B | 18 months follow up
  A simple measure of executive cognitive function
DS-14 | 18 months follow up
  A standard assessment of negative affectivity, social inhibition, and type D personality, which might be related to poor cardiovascular prognosis.

OTHER OUTCOMES:
VO2-peak | 18 months follow up
  VO2-peak is obtained by use of a symptom limited treadmill test to measure cardiovascular fitness.
  This measure is only used in the Trondheim arm of the study

CONTACTS AND LOCATIONS:
Overall Officials: Bent Indredavik, Prof, Study Director — National Taiwan Normal University; Torunn Askim, PhD, Principal Investigator — National Taiwan Normal University
Locations (2):
- Norway (2):
  - Bærum Hospital, Sandvika
  - St. Olavs Hospital, Trondheim

REFERENCES:
- [Background] Askim T, Langhammer B, Ihle-Hansen H, Magnussen J, Engstad T, Indredavik B. A Long-Term Follow-Up Programme for Maintenance of Motor Function after Stroke: Protocol of the life after Stroke-The LAST Study. Stroke Res Treat. 2012;2012:392101. doi: 10.1155/2012/392101. Epub 2012 Nov 22. PMID 23227428
- [Result] Askim T, Langhammer B, Ihle-Hansen H, Gunnes M, Lydersen S, Indredavik B; LAST Collaboration Group. Efficacy and Safety of Individualized Coaching After Stroke: the LAST Study (Life After Stroke): A Pragmatic Randomized Controlled Trial. Stroke. 2018 Feb;49(2):426-432. doi: 10.1161/STROKEAHA.117.018827. Epub 2017 Dec 28. PMID 29284737
- [Result] Dohl O, Halsteinli V, Askim T, Gunnes M, Ihle-Hansen H, Indredavik B, Langhammer B, Phan A, Magnussen J. Factors contributing to post-stroke health care utilization and costs, secondary results from the life after stroke (LAST) study. BMC Health Serv Res. 2020 Apr 6;20(1):288. doi: 10.1186/s12913-020-05158-w. PMID 32252739
- [Derived] Saunders DH, Mead GE, Fitzsimons C, Kelly P, van Wijck F, Verschuren O, Backx K, English C. Interventions for reducing sedentary behaviour in people with stroke. Cochrane Database Syst Rev. 2021 Jun 29;6(6):CD012996. doi: 10.1002/14651858.CD012996.pub2. PMID 34184251
- [Derived] Gunnes M, Indredavik B, Langhammer B, Lydersen S, Ihle-Hansen H, Dahl AE, Askim T; LAST Collaboration group. Associations Between Adherence to the Physical Activity and Exercise Program Applied in the LAST Study and Functional Recovery After Stroke. Arch Phys Med Rehabil. 2019 Dec;100(12):2251-2259. doi: 10.1016/j.apmr.2019.04.023. Epub 2019 Jul 30. PMID 31374191